CLINICAL TRIAL: NCT06770374
Title: Effectiveness of a Zinc Oxide Adhesive Securement Device in the Fixation of Midline and Peripherally Inserted Central Catheters in Hospitalized Adult Patients: Randomised Clinical Trial
Brief Title: Effectiveness of a Zinc Oxide Adhesive Securement Device in the Fixation of Midline and Peripherally Inserted Central Catheters in Hospitalized Adult Patients
Acronym: FIX-ETI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Arnau de Vilanova (Other)
Collaborators: Official College of Nurses of Lleida (Unknown); Catalan Institute of Health (Other Government)
Responsible Party: Principal Investigator, Ferran Padilla Nula, Principal Investigator, Hospital Arnau de Vilanova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03/24
Record Dates: First submitted 2024-12-24; First posted 2025-01-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Vascular Access Complication; Skin and Subcutaneous Tissue Disorders; Phlebitis; Pain
Keywords: Catheters; Vascular Access Devices; Catheter-Related Infections; Nurse Specialists; Nurses; Randomised Controlled Trial
MeSH Terms: conditions — Skin Diseases; Phlebitis; Pain; Catheter-Related Infections | interventions — Methods; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Classic parallel model with an intervention group, where the catheters will be fixed with a zinc oxide fixation dressing (Grip-Lok® Ref.2200NUZA), and a control group where the catheters will be fixed with a dressing without zinc oxide (acrylic adhesive) (Grip-Lok® Ref.3300MWA).
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers are the ones who performed the insertion of the catheters and the subsequent data collection, but the patients do not know which ones have the zinc oxide device and which ones do not. In addition, the results will be evaluated by a researcher external to the data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): After cannulation of a midline or peripherally inserted central venous catheter with modified micro-Seldinger technique, the control group underwent standard care.
  Interventions: Procedure: Control group: acrylic adhesive sutureless fixation device; Device: PICC; Device: Midline; Other: Ultrasound scanner
- Intervention (Experimental): After cannulation of a midline or peripherally inserted central venous catheter with modified micro-Seldinger technique, the intervention group underwent the alternative care.
  Interventions: Procedure: Intervention Group: zinc oxide sutureless fixation device; Device: PICC; Device: Midline; Other: Ultrasound scanner

INTERVENTIONS:
Procedure: Control group: acrylic adhesive sutureless fixation device — The standard care consists of:
  * Application of hemostasis at the point of insertion for 2 minutes post puncture or until bleeding stops.
  * Fix with clear polyurethane dressing (3M®-1655 Tegaderm™ IV), cyanoacrylate glue (SecurePortIV®) and acrylic adhesive sutureless fixation device (3300MWA Grip-Lok®).
  Other Names: Control
  Arms: Control
Procedure: Intervention Group: zinc oxide sutureless fixation device — Alternative care consisted of:
  * Application of haemostasis at the insertion site for 2 minutes post-puncture or until cessation of bleeding.
  * Fixation with clear polyurethane dressing (3M®-1655 Tegaderm™ IV), cyanoacrylate glue (SecurePortIV®) and zinc oxide sutureless fixation device (2200NUZA Grip-Lok®).
  Other Names: Intervention
  Arms: Intervention
Device: PICC — The PICC lines used in the study will all be third-generation polyurethane and of the commercial brands:
  * PowerPICC™ 4, 5 and 6 Fr from BD
  * Maxflo expert™ 5 and 6 Fr from Vygon
Device: Midline — The midline lines used in the study will be second or third generation polyurethane and of the commercial brands:
  * PowerMidline™ 4 Fr from BD
  * Arrow® Midline 4Fr from Arrow
Other: Ultrasound scanner — All punctures will be performed under ultrasound guidance.
  Other Names: Ultrasound

SUMMARY:
Study in which a zinc oxide fixation device (a product that can help protect the skin) for catheters (polyurethane tubes inserted into a vein) will be tested to reduce catheter-related complications: catheter displacement, skin complications, phlebitis and pain..

DETAILED DESCRIPTION:
Introduction: Midline catheters (MLC) and peripherally inserted central catheters (PICC) are commonly used vascular access devices (VAD) in healthcare institutions where infusion therapies are required, and have been proven to have an optimal level of safety and efficacy for intravenous drug delivery. However, the insertion of these VADs has a number of potential associated complications (immediate, early and/or late), and proper fixation may reduce them.

Hypothesis: Using a zinc oxide adhesive securement device (ASD) reduces the number of fixation-associated complications in MLC and PICC compared to a universal ASD with silicone adhesive.

Objective: To evaluate the efficacy of using a ASD with zinc oxide for post insertion fixation of MLC and PICC in hospitalised adult patients.

Methodology: Randomised clinical study. Two randomised groups will be created before catheter cannulation. The control group will be cured with an ASD with acrylic adhesive (Grip-Lok® Ref.3300MWA) and the intervention group will be cured with ASD with zinc oxide (Grip-Lok® Ref.2200NUZA).

Expected results: The investigators expect to reduce the number of complications related to the attachment of PICCs and MLCs in adult hospitalised patients following the protocolised placement of a ASD with zinc oxide during the first cure. Specifically, it is expected to reduce the number of catheter dislodgements, the number of medical adhesive-related skin injuries (MARSI) and the amount of phlebitis.

Clinical implication: The study will help to improve decision making related to maintenance and care of VAD in order to reduce the main associated complications.

ELIGIBILITY:
Inclusion Criteria:

* requiring cannulation of a midline catheter or a PICC
* who accepted and signed the informed consent voluntarily
* with an inpatient unit admission of minimum 7 days

Exclusion Criteria:

- patients with a known allergy to zinc oxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 7 days
  Percentage of participants with adverse events following cannulation of a midline or peripherally inserted central catheter after fixation with a zinc oxide sutureless fixation device.

SECONDARY OUTCOMES:
Number of participants with altered skin under the sutureless fixation device assessed by observation (yes/no). | 7 days
  Percentage of participants with skin alterations under the sutureless fixation device after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four examinations will be performed: post puncture, at 24 hours, at 72 hours and at 7 days, in which the puncture site will be visualized for signs of skin alterations and it will be noted whether they exist and what type (Hematoma, Skin Stripping, Tension Injury or Blister, Skin Tear, Irritant Contact Dermatitis, Allergic Contact Dermatitis, Maceration or Folliculitis).
Number of participants with post-treatment catheter displacement assessed by observation (yes/no). | 7 days
  Percentage of participants with catheter displacement after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the puncture site will be visualized to check if the catheter is still in the same point or if it has been displaced.
Number of participants with post-treatment phlebitis assessed with the Maddox visual phlebitis rating scale. | 7 days
  Percentage of participants with phlebitis after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the puncture site will be visualized to check for signs of phlebitis, according to the Maddox scale.
Number of participants with post-treatment pain in extremity assessed with the EVA scale. | 7 days
  Percentage of participants with pain in extremity after puncture of a midline or central venous catheter with the modified micro-Seldinger technique. Four cures will be performed: post puncture, at 24 hours, 72 hours and 7 days, where the patient will be asked what pain he/she feels in the extremity related to the catheter.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Arnau de Vilanova Hospital, Lleida, Catalonia
  - Hospital Universitari Arnau de Vilanova, Lleida, Catalonia

IPD SHARING:
Plan to Share IPD: Yes
The data from the FIX-ETI project were uploaded to Mendelay data, so that the data can be observed and analyzed by the entire scientific community and anyone interested in the subject.
  The research protocol, the informed consent, the infographic presented to the patients, the data collection notebook and the data collected during all the cures will be uploaded and retrieved from the REDCap database.
Supporting Information: Study Protocol, ICF
Time Frame: They will be available by the end of 2025.
Access Criteria: Will be accessible to everyone through the Mendelay data platform.
URL: https://data.mendeley.com/preview/bjj9kz5ntw

REFERENCES:
- [Background] Huskisson EC, Jones J, Scott PJ. Application of visual-analogue scales to the measurement of functional capacity. Rheumatol Rehabil. 1976 Aug;15(3):185-7. doi: 10.1093/rheumatology/15.3.185. PMID 968347
- [Background] Babaieasl F, Yarandi HN, Saeidzadeh S, Kheradmand M. Comparison of EMLA and Diclofenac on Reduction of Pain and Phlebitis Caused by Peripheral IV Catheter: A Randomized-Controlled Trial Study. Home Healthc Now. 2019 Jan/Feb;37(1):17-22. doi: 10.1097/NHH.0000000000000704. PMID 30608463
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Lansdown AB, Mirastschijski U, Stubbs N, Scanlon E, Agren MS. Zinc in wound healing: theoretical, experimental, and clinical aspects. Wound Repair Regen. 2007 Jan-Feb;15(1):2-16. doi: 10.1111/j.1524-475X.2006.00179.x. PMID 17244314
- [Background] Kogan S, Sood A, Garnick MS. Zinc and Wound Healing: A Review of Zinc Physiology and Clinical Applications. Wounds. 2017 Apr;29(4):102-106. PMID 28448263
- [Background] Molina-Mazon CS, Martin-Cerezo X, Domene-Nieves de la Vega G, Asensio-Flores S, Adamuz-Tomas J. Comparative study on fixation of central venous catheter by suture versus adhesive device. Enferm Intensiva (Engl Ed). 2018 Jul-Sep;29(3):103-112. doi: 10.1016/j.enfi.2017.10.004. Epub 2018 Mar 27. English, Spanish. PMID 29602709
- [Background] Xu H, Hyun A, Mihala G, Rickard CM, Cooke ML, Lin F, Mitchell M, Ullman AJ. The effectiveness of dressings and securement devices to prevent central venous catheter-associated complications: A systematic review and meta-analysis. Int J Nurs Stud. 2024 Jan;149:104620. doi: 10.1016/j.ijnurstu.2023.104620. Epub 2023 Oct 9. PMID 37879273
- [Background] Bing S, Smotherman C, Rodriguez RG, Skarupa DJ, Ra JH, Crandall ML. PICC versus midlines: Comparison of peripherally inserted central catheters and midline catheters with respect to incidence of thromboembolic and infectious complications. Am J Surg. 2022 May;223(5):983-987. doi: 10.1016/j.amjsurg.2021.09.029. Epub 2021 Sep 25. PMID 34600737
- [Background] Moureau N, Chopra V. Indications for peripheral, midline and central catheters: summary of the MAGIC recommendations. Br J Nurs. 2016 Apr 28-May 11;25(8):S15-24. doi: 10.12968/bjon.2016.25.8.S15. PMID 27126759
- [Background] Woller SC, Stevens SM, Evans RS. The Michigan Appropriateness Guide for Intravenous Catheters (MAGIC) initiative: A summary and review of peripherally inserted central catheter and venous catheter appropriate use. J Hosp Med. 2016 Apr;11(4):306-10. doi: 10.1002/jhm.2525. Epub 2015 Dec 14. PMID 26662622
- [Background] Chan RJ, Northfield S, Larsen E, Mihala G, Ullman A, Hancock P, Marsh N, Gavin N, Wyld D, Allworth A, Russell E, Choudhury MA, Flynn J, Rickard CM. Central venous Access device SeCurement And Dressing Effectiveness for peripherally inserted central catheters in adult acute hospital patients (CASCADE): a pilot randomised controlled trial. Trials. 2017 Oct 4;18(1):458. doi: 10.1186/s13063-017-2207-x. PMID 28978332
- [Background] Gravdahl E, Steine S, Augestad KM, Fredheim OM. Use and safety of peripherally inserted central catheters and midline catheters in palliative care cancer patients: a retrospective review. Support Care Cancer. 2023 Sep 19;31(10):580. doi: 10.1007/s00520-023-08045-2. PMID 37725150
- [Background] Kleidon TM, Schults JA, Wainwright C, Mihala G, Gibson V, Saiyed M, Byrnes J, Cattanach P, Macfarlane F, Graham N, Shevill E, Ullman AJ. Comparison of midline catheters and peripherally inserted central catheters to reduce the need for general anesthesia in children with respiratory disease: A feasibility randomized controlled trial. Paediatr Anaesth. 2021 Sep;31(9):985-995. doi: 10.1111/pan.14229. Epub 2021 Jun 21. PMID 34053159
- [Background] Thomsen SL, Boa R, Vinter-Jensen L, Rasmussen BS. Safety and Efficacy of Midline vs Peripherally Inserted Central Catheters Among Adults Receiving IV Therapy: A Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2355716. doi: 10.1001/jamanetworkopen.2023.55716. PMID 38349655
- [Background] Urtecho M, Torres Roldan VD, Nayfeh T, Espinoza Suarez NR, Ranganath N, Sampathkumar P, Chopra V, Safdar N, Prokop LJ, O'Horo JC. Comparing Complication Rates of Midline Catheter vs Peripherally Inserted Central Catheter. A Systematic Review and Meta-analysis. Open Forum Infect Dis. 2023 Jan 18;10(2):ofad024. doi: 10.1093/ofid/ofad024. eCollection 2023 Feb. PMID 36751645
- [Background] Nickel B, Gorski L, Kleidon T, Kyes A, DeVries M, Keogh S, Meyer B, Sarver MJ, Crickman R, Ong J, Clare S, Hagle ME. Infusion Therapy Standards of Practice, 9th Edition. J Infus Nurs. 2024 Jan-Feb 01;47(1S Suppl 1):S1-S285. doi: 10.1097/NAN.0000000000000532. No abstract available. PMID 38211609
- [Result] Padilla-Nula F, Bergua-Lorente A, Farrero-Mena J, Escola-Nogues A, Llaurado-Mateu M, Serret-Nuevo C, Bellon F. Effectiveness of cyanoacrylate glue in the fixation of midline catheters and peripherally inserted central catheters in hospitalised adult patients: Randomised clinical trial (CIANO-ETI). SAGE Open Med. 2023 Apr 28;11:20503121231170743. doi: 10.1177/20503121231170743. eCollection 2023. PMID 37152837